CLINICAL TRIAL: NCT01309152
Title: Peri-and Postoperative Subcutaneous Adipose Tissue Cefazolin Determination Using Microdialysis in Morbidly Obese and Non-obese Patients
Brief Title: Cefazolin Subcutaneous Microdialysis in Morbidly Obese Patients
Acronym: MICK
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: CAJ Knibbe, St. Antonius Hospital
Other Study IDs: MICK R-10.29A/MICK; LTME/VL-10.14/MICK
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Morbid Obesity
Keywords: cefazolin; microdialysis; morbid obesity; pharmacokinetics
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and microdialysis filtrate of subcutenous tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that cefazolin perfusion to subcutaneous adipose tissue is reduced in morbidly obese patients. The primary objective of this exploratory pilot study is therefore to investigate target site (subcutaneous adipose tissue) penetration of cefazolin in morbidly obese patients and non-obese patients. The investigators aim to examine whether and how cefazolin plasma concentrations are predictive of subcutaneous (target) cefazolin concentrations. Possible factors of influence on the distribution of cefazolin (tissue perfusion, body weight, distribution of adipose tissue, other) will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index > 40 kg/m2
* BMI between 20-25
* undergoing laparoscopic gastric banding, or bypass surgery or sleeve gastrectomy (See population description for surgery type of the non-obese group)
* 21-60 years old
* American Society of Anaesthesiologists (ASA) physical status II to III

Exclusion Criteria:

* pregnancy
* breastfeeding
* known allergy for cefazolin/nadroparin
* known ejection fraction of < 35%
* renal insufficiency

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 8 morbidly obese patients undergoing weight reducing surgery And 8 non-obese patients undergoing surgery which will require an arterial line, nadroparin and cefazolin administration perioperatively and postoperative stay at the Post-Anesthesia Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - St Antonius Hospital, Nieuwegein, Utrecht
  - St Antonius Hospital, Nieuwegein
  - St. antonius hospital, Nieuwegein

REFERENCES:
- [Derived] Diepstraten J, Janssen EJ, Hackeng CM, van Dongen EP, Wiezer RJ, van Ramshorst B, Knibbe CA. Population pharmacodynamic model for low molecular weight heparin nadroparin in morbidly obese and non-obese patients using anti-Xa levels as endpoint. Eur J Clin Pharmacol. 2015 Jan;71(1):25-34. doi: 10.1007/s00228-014-1760-4. Epub 2014 Oct 12. PMID 25304008
- [Derived] Brill MJ, Houwink AP, Schmidt S, Van Dongen EP, Hazebroek EJ, van Ramshorst B, Deneer VH, Mouton JW, Knibbe CA. Reduced subcutaneous tissue distribution of cefazolin in morbidly obese versus non-obese patients determined using clinical microdialysis. J Antimicrob Chemother. 2014 Mar;69(3):715-23. doi: 10.1093/jac/dkt444. Epub 2013 Nov 8. PMID 24214905